CLINICAL TRIAL: NCT05770063
Title: Effect of Compound Amino Acid Tablets on Nutritional Status of Patients With Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Chest Hospital (Other)
Responsible Party: Principal Investigator, Zhuo Li, Beijing Chest Hospital, Beijing Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: YNLX-2022-011
Record Dates: First submitted 2023-02-21; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Amino Acid Deficiency; Malnutrition; Lung Cancer
MeSH Terms: conditions — Malnutrition; Lung Neoplasms | interventions — Amino Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): compound amino acid supplement
  Interventions: Dietary Supplement: amino acid tablet
- control group (Placebo Comparator): placebo
  Interventions: Dietary Supplement: amino acid tablet

INTERVENTIONS:
Dietary Supplement: amino acid tablet — multiple essential amino acids supplements

SUMMARY:
To investigate whether compound amino acid supplementation can further promote protein synthesis and improve nutritional status for lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* NRS2002 >=3 scores
* lung cancer patients
* low albumin or hemoglobin
* informed consent

Exclusion Criteria:

* Acute and critical patients;
* Severe liver and kidney dysfunction;
* Patients with gastrointestinal bleeding or intestinal obstruction;
* Pregnant women, lactating women, people with mental illness, and people without independent behavior ability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-04-15 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Concentration of albumin | after 42 days after the intervention